CLINICAL TRIAL: NCT07250074
Title: "Sentinella" Project: a Digital Registry and Education Network for Child Maltreatment Protection.
Brief Title: "Sentinella": Registry and Training for Child Protection
Acronym: Sentinella
Status: Not yet recruiting | Type: Observational
Sponsor: Buzzi Children's Hospital (Other)
Responsible Party: Principal Investigator, Valeria Calcaterra, Prof, Buzzi Children's Hospital
Other Study IDs: Buzzi021125
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Child Abuse; Child Neglect; Child Maltreatment

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Integrated Digital Registry and Education Intervention — The Sentinella intervention combines a secure digital registry with a structured training program for healthcare professionals to improve the early recognition and reporting of suspected child maltreatment. The digital registry, developed using the REDCap platform, enables standardized, anonymous data collection and supports communication between hospital and community services. The training component includes theoretical and practical modules focused on clinical, psychological, and legal aspects of child abuse, as well as hands-on exercises for correct use of the registry.
  This integrated approach-linking technology and professional education-distinguishes Sentinella from other interventions, which typically address either training or data collection separately.

SUMMARY:
The "Sentinella" project aims to improve the early recognition and prevention of child maltreatment by creating a digital registry and education network for healthcare professionals. The study will test a new online registry built on the REDCap platform to collect standardized, anonymous data about suspected cases of abuse or neglect. It also includes a structured training program for pediatricians and other healthcare workers to strengthen their skills in identifying and reporting maltreatment.

This observational study will assess how easy the registry is to use and whether the training improves participants' knowledge and reporting practices. The project is expected to enhance collaboration between hospitals and community services, reduce reporting delays, and create a model for regional or national systems to protect vulnerable children.

DETAILED DESCRIPTION:
Child maltreatment is a major public health concern that affects one billion children worldwide each year. In Italy, despite legislative progress, the detection and reporting of suspected cases remain fragmented, often due to lack of standardized systems and professional training.

The Sentinella project aims to address these gaps by integrating a digital registry for the anonymous reporting of suspected child maltreatment with a structured training program for healthcare professionals. The project combines technological innovation and education to strengthen early recognition, documentation, and reporting within the pediatric network.

The study is observational, exploratory, and monocentric, lasting 24 months. It includes two main components:

1. Registry Phase: Development and evaluation of a secure digital registry based on the REDCap platform for standardized and anonymous data collection. Usability is measured with the System Usability Scale (SUS), where a score ≥70 indicates good usability and ≥80 excellent usability.
2. Training Phase: A blended theoretical and practical course (approximately 20 hours) addressing clinical, psychological, and legal aspects of child abuse, communication skills, and proper use of the registry. Training effectiveness is measured through pre- and post-tests and participant satisfaction questionnaires.

The target population consists of approximately 30 healthcare professionals (pediatricians, psychologists, nurses, and social workers) who voluntarily participate, complete the training, and consent to data collection. No patient data are collected, and no clinical interventions are performed.

Primary outcome: Usability of the digital registry (SUS score). Secondary outcomes: Improvement in knowledge and competence, increased reporting rates, and user satisfaction.

Data will be analyzed using descriptive and inferential statistics (paired t-tests, Wilcoxon tests, Poisson or negative binomial regression models). Significance will be set at p < 0.05.

The project complies with the Declaration of Helsinki and the EU GDPR (Reg. 2016/679). Participation is voluntary and risk-free.

Expected results: The registry is expected to achieve high usability (SUS ≥80), while the training program should lead to measurable improvement in professional knowledge and reporting behavior. Together, these components aim to enhance coordination between hospital and community services, increase early detection of abuse, and establish a sustainable "Sentinel Pediatricians" network.

Ultimately, Sentinella seeks to validate an integrated and replicable model for child protection that can evolve into an Observatory on Child Maltreatment, supporting continuous surveillance, education, and policy development.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals (e.g., pediatricians, psychologists, nurses, social workers) working within the regional pediatric network.
* Voluntary participation in the Sentinella project.
* Completion of the planned training program (theoretical and practical components).
* Willingness to use the digital registry and complete evaluation questionnaires.
* Provision of written informed consent.

Exclusion Criteria:

* Failure to complete the full training program.
* Partial participation in simulation or practical sessions.
* Incomplete pre- and post-training questionnaires.
* Refusal or withdrawal of informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of healthcare professionals involved in child care and protection within the regional pediatric network, including hospital and community pediatricians, psychologists, nurses, and social workers. Participants are professionals who voluntarily enroll in the Sentinella project, complete the structured training program, and participate in the evaluation of the digital registry's usability and the training's effectiveness.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-12-03 (Estimated); Primary Completion 2026-05-03 (Estimated); Study Completion 2027-11-03 (Estimated)

PRIMARY OUTCOMES:
System Usability of the Digital Registry | At the end of the registry implementation phase (approximately 6 months after activation).
  Evaluation of the usability and acceptability of the Sentinella digital registry among participating healthcare professionals, measured using the System Usability Scale (SUS). The SUS provides a standardized usability score ranging from 0 to 100; a score ≥70 indicates good usability, and ≥80 indicates excellent usability.

IPD SHARING:
Plan to Share IPD: No